CLINICAL TRIAL: NCT05067712
Title: Treatment of Palatally Displaced Maxillary Canines - a Controlled Randomized Clinical Trial
Brief Title: The Effect of Surgical Technique on PDC
Acronym: PDC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Jonkoping County Hospital (Other)
Responsible Party: Principal Investigator, Lucete Fernandes faerovig, Principal investigator, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015715
Record Dates: First submitted 2021-06-03; First posted 2021-10-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Embedded and Impacted Teeth
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Surgical Exposure Technique (Active Comparator): After randomization, the PDC allocated to this arm is surgically exposed with the Open Technique followed by the Orthodontic Treatment phase
  Interventions: Procedure: Open Surgical Exposure Technique
- Closed Surgical Exposure Technique (Active Comparator): After randomization, the PDC allocated to this arm is surgically exposure with the Closed technique followed by the Orthodontic Treatment phase.
  Interventions: Procedure: Closed Surgical Exposure Technique

INTERVENTIONS:
Procedure: Open Surgical Exposure Technique — * A mucoperiosteal palatal flap is elevated off the bone from the premolar to the midline
  * The bone covering the crown aspect of the canine is removed until the largest diameter of the crown is exposed
  * Follicular tissue is removed from the exposed crown area
  * The flap is repositioned back and sutured
  * The area over the exposed canine crown is excised leaving a window with the crown uncovered.
  * If the tooth is deeply embedded in the bone, a dressing is placed over the uncovered crown and kept in place with sutures.
  * The extraction of the primary canine (if present) is made before or in connection with the surgical exposure.
  * Ten to fifteen days later the dressing and sutures are removed and the tooth is left to erupt autonomously.
  * When the canine has spontaneously erupted above the palatal mucosa an attachment is bonded to the crown and the canine is moved into alignment in the dental arch above the mucosa with orthodontic appliances.
  Arms: Open Surgical Exposure Technique
Procedure: Closed Surgical Exposure Technique — * A mucoperiosteal palatal flap is elevated off the bone from the premolar to the midline
  * The bone covering the crown aspect of the canine is removed until the largest diameter of the crown is exposed.
  * Follicular tissue is removed from the exposed crown area.
  * An attachment with a chain is bonded to the exposed canine crown.
  * The flap is repositioned back and sutured to cover the exposed crown leaving the chain through the palatal mucosa free in the oral cavity
  * The extraction of the primary canine (if present) made before or in connection with the surgical exposure
  * Ten to fifteen days later the sutures are removed.
  * Within days, traction is applied to the canine with orthodontic appliances by means of the chain, and the canine is pulled through the palatal mucosa out to the oral cavity and into alignment in the dental arch.
  Arms: Closed Surgical Exposure Technique

SUMMARY:
Permanent maxillary canines are the second teeth that most commonly assume ectopic positions after the third molars. They are diagnosed as impacted and have an incidence of 1 % to 3%

In their ectopic path of eruption, they can cause damage (resorption) of the adjacent roots, a severe complication that may lead to the loss of anterior teeth. When cone-beam computed tomography (CT) scanning is used for diagnose, root resorption is detected in two-thirds of the lateral incisors adjacent to impacted maxillary canines before treatment.

The treatment of this condition comprises two stages: a surgical intervention to uncover the canine crown followed by orthodontic treatment to move the canine into correct position. The surgical intervention commonly involves two different techniques: the open and the closed technique.

The open technique procedure involves removing the bone and mucosa covering the crown of the canine. The exposed crown is left uncovered and a pack is placed over the area to avoid overgrowth of tissue. When enough spontaneous eruption of the canine has occurred, an orthodontic attachment is bonded to the crown and the tooth is moved above the mucosa with orthodontic appliances into the correct position.

The closed technique procedure involves bonding an orthodontic attachment to the crown with a chain after exposing the canine during the surgery. The palatal flap is sutured back covering the exposed crown and the chain is left through the palatal mucosa free in the oral cavity. Shortly after, the canine is forced to erupt through the palatal mucosa and moved into the correct position with orthodontic appliances.

The purpose of this prospective randomized clinical trial is to compare outcome variables between the Open and Closed surgical exposure techniques regarding the success of treatment, patient's perceptions of pain and discomfort experienced and analgesic consumption, treatment time, and complications. The null hypothesis is that similar outcomes occur when the surgical exposure of palatally impacted canines is performed by using the open or the closed surgical technique.

DETAILED DESCRIPTION:
Consecutive patients planned for surgical exposure of uni- or bilateral palatally impacted canines of two centers, are invited to participate in the Trial. The centers are the University Orthodontic Departments of Oslo, Norway, and Jonkoping, Sweden.

Potential participant patients and their parents are given verbal and written information about the Trial and Informed Consent is obtained.

Participants are randomly allocated to one of two interventions by use of Permuted Block Randomization in order to maintain equal allocations across treatment groups. Allocation concealment is held by one individual in each center that is not involved in the study. No stratification is made for age or gender in the two groups.

If the maxillary deciduous canine is present at the time of the surgery, the tooth is removed together with the exposure of the impacted canine.

Before entering the surgery room, participants answer a first questionnaire on whether they are experiencing pain or discomfort (measured in VAS-scales) in the area of the impacted canine and whether they have taken analgesics. The questionnaire is filled in and delivered back before entering the surgery room. After the surgical exposure, verbal and written information and recommendations on chlorhexidine mouth rinse and analgesic consumption are given. A second questionnaire is then handed out for participants to self-report the pain-discomfort they experienced during surgery, and are experiencing in the evening the same day and the following seven days together with the analgesic consumption. The second questionnaire is delivered back to the clinic at the post-surgical control.

At the post-surgical control, participants receive a third questionnaire where they self-report the pain-discomfort they experienced during and after sutures (closed technique) and packing (open technique) are removed.

After the surgical exposure with the open technique, the canine is left to erupt spontaneously. Participants are follow-up by the orthodontist until the canine has erupted enough (approximately ½ - 1/3 of the crown above the level of the palatal mucosa) to bond an attachment to the crown. The canine then starts to be moved into alignment in the dental arch above the mucosa with orthodontic appliances.

After the surgical exposure with the closed technique, the impacted canine starts to be moved with orthodontic appliances within 2 weeks after surgery. The canine is moved into alignment in the dental arch through the mucosa.

From the completion of the surgical exposure phase until the previously impacted canine is orthodontically positioned in the dental arch, similar questionnaires are handed out to the participants in both treatment groups every second/ third orthodontic control.

The participants are followed until the active orthodontic treatment is finished and orthodontic retainers bonded.

Schedule/ registrations:

Before the surgical exposure phase of treatment (T0)

* Clinical anamnesis
* Routine dental clinical examination. Assessment of periodontal pocket depth, gingival bleeding on probing, gingival recession in the lateral incisor in the impacted and nonimpacted contralateral side.
* Study models. Assessment of occlusion traits, presence of maxillary deciduous canine.
* Panoramic radiograph. Assessment of the position of the impacted canine: mesial position, mesial inclination, and distance to the occlusal line according to Ericson and Kurol.
* Cephalogram. Assessment of upper incisor sagittal inclination.
* CBCT (cone beam computed tomography). Assessment of the exact impacted canine position, size of the impacted canine's follicle, crestal bone height in the lateral incisor in the impacted and nonimpacted contra lateral side, root resorption of the impacted canine, lateral incisor, and first premolar in the impacted and nonimpacted contra lateral side

Surgical exposure day (T1)

* Questionnaires are handed out to the participants for assessment of pain and discomfort (measured on VAS-scale) and analgesic consumption : (1) before surgery same day (2) after surgery same day and following 7 days, (3) post-surgery control same day and following 7 days.
* Registrations at the surgery: duration of the operation, complications, depth of the impacted canine from the mucosa surface.

The previously palatally impacted canine has erupted (approximately 1/3-1/2 canine crown above palatal mucosa) (T2)

* Questionnaires are handed out to participants between T1 and T2 for assessment of pain and discomfort (measured on VAS-scale) and analgesic consumption the same day and following 7 days after every second/ third orthodontic control
* Timespan T1-T2
* Complications associated with the eruption of the canine since surgery

The previously palatally impacted canine is aligned in the dental arch and ligated to a 0.016 X 0.022 nickel-titanium / standard steel archwire in the 0.018- appliance system or a 0.019 X 0.025 nickel-titanium / standard steed archwire in the 0.022- appliance system (T3)

* CBCT (cone beam computed tomography). Assessment of the position of the canine root, crestal bone height in the canine, lateral incisor, and first premolar in the impacted and nonimpacted contra lateral side, root resorption of the impacted canine, incisors, and first premolar in the impacted and nonimpacted contra lateral side
* Questionnaires are handed out to participants between T2 and T3 for assessment of pain and discomfort (measured on VAS-scale) and analgesic consumption the same day and following 7 days after every second/ third orthodontic control
* Timespan T2-T3
* Complications associated with the orthodontic alignment of the previously impacted canine into the dental arch.

The active orthodontic treatment is finished and an orthodontic retainer is fitted (T4)

* Routine clinical examination. Assessment of periodontal pocket depth, gingival bleeding on probing, gingival recession in the canine, incisors and first premolar in the impacted and nonimpacted contra lateral side.
* Study models. Assessment of occlusion traits.
* Panoramic radiograph. Assessment of root parallelism, root resorption.
* Cephalogram. Assessment of upper incisor sagittal inclination.

Except for the CBCT examinations and questionnaires, all the examinations and treatments performed in this trial are the routine examinations and treatments of palatally impacted maxillary canines performed in Norway and Sweeden. All the surgical exposures and orthodontic treatments are performed by or under the supervision of the same specialist in oral surgery and orthodontics, respectively, in each center, with many years of experience.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients diagnosed with palatally impacted canine with a sagittal position in Zone 2-4 as documented on panoramic radiographs according to the criteria proposed by Ericson and Kurol,1988, planned to start treatment with surgical exposure of the impacted canine.
* Patients with uni- or bilateral impacted canines are included. In bilateral impaction cases, the more severely positioned impacted canine according to the Zone (Zone 2 - 4) is included in the trial.
* No restriction of presenting malocclusion
* Dental developmental stage: Maxillary DS2M1 and DS3M2 according to Bjork.
* Age not older than 16 years at surgery

Exclusion Criteria:

* Agenesis of lateral incisors on the impaction side
* Peg-shaped lateral incisors on the impaction side
* Previous orthodontic treatment
* Subjects with craniofacial deformity/ syndromes
* Documented learning disability
* Communication problems related to the language when an interpreter is needed
* Sagittal position of the impacted canine in Zone 5, according to Ericson and Kurol, documented on panoramic radiographs.

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Success of treatment | Within 3 years from surgery
  The canine is aligned in the dental arch. "Aligned in the dental arch" meaning the canine being ligated to a 0.016 X .0.22 nickel- titanium/ standard steel in a 0.018-appliance system or to a 0.019 X 0.025 nickel-titanium/ standard steel arch-wire in a 0.022- appliance system
Patient's perceptions of pain-discomfort experience and analgesic consumption | Within 3 years from surgery
  Perceptions of pain-discomfort experienced and analgesic consumption are self reported on a 100 mm visual analogue scale (VAS) and questionnaires in the first evening and the following 7 evenings, after surgery, after suture and pack removal and after every second/ third orthodontic activation.

SECONDARY OUTCOMES:
Canine eruption time | Within 1,5 years from surgery
  Time span from the surgery until 1/3 to 1/2 of the canine crown is above the level of the palatal mucosa

OTHER OUTCOMES:
Surgery operation time | 1,5 hours
  Time span (hours, minutes) from the first incision to the last suture
Complications associated with the surgical technique | Within 1,5 years from the surgery
  Presence, number and type of complications associated with the surgery
Duration of orthodontic treatment | Within 3 years from the surgery
  Time span from surgery until the canine being ligated to a 0.016 X 0.022 nickel-titanium/

CONTACTS AND LOCATIONS:
Overall Officials: Lucete Fe Færøvig, Principal Investigator — University of Oslo
Locations (2):
- Det Odontologiske Fakultet, avdelingen for kjeveortopedi, Oslo, Norway
- Odontologiska Institutionen, avdelingen för ortodonti, Jönköping, Sweden

REFERENCES:
- [Background] Ericson S, Kurol J. Radiographic examination of ectopically erupting maxillary canines. Am J Orthod Dentofacial Orthop. 1987 Jun;91(6):483-92. doi: 10.1016/0889-5406(87)90005-9. PMID 3473928
- [Background] Bishara SE. Impacted maxillary canines: a review. Am J Orthod Dentofacial Orthop. 1992 Feb;101(2):159-71. doi: 10.1016/0889-5406(92)70008-X. PMID 1739070
- [Background] Peck S, Peck L, Kataja M. The palatally displaced canine as a dental anomaly of genetic origin. Angle Orthod. 1994;64(4):249-56. doi: 10.1043/0003-3219(1994)0642.0.CO;2. PMID 7978519
- [Background] Walker L, Enciso R, Mah J. Three-dimensional localization of maxillary canines with cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2005 Oct;128(4):418-23. doi: 10.1016/j.ajodo.2004.04.033. PMID 16214621
- [Background] Stewart JA, Heo G, Glover KE, Williamson PC, Lam EW, Major PW. Factors that relate to treatment duration for patients with palatally impacted maxillary canines. Am J Orthod Dentofacial Orthop. 2001 Mar;119(3):216-25. doi: 10.1067/mod.2001.110989. PMID 11244415
- [Background] Spencer HR, Ramsey R, Ponduri S, Brennan PA. Exposure of unerupted palatal canines: a survey of current practice in the United Kingdom, and experience of a gingival-sparing procedure. Br J Oral Maxillofac Surg. 2010 Dec;48(8):641-4. doi: 10.1016/j.bjoms.2009.08.032. Epub 2009 Nov 3. PMID 19889488
- [Background] Pearson MH, Robinson SN, Reed R, Birnie DJ, Zaki GA. Management of palatally impacted canines: the findings of a collaborative study. Eur J Orthod. 1997 Oct;19(5):511-5. doi: 10.1093/ejo/19.5.511. PMID 9386337
- [Background] Counihan K, Al-Awadhi EA, Butler J. Guidelines for the assessment of the impacted maxillary canine. Dent Update. 2013 Nov;40(9):770-2, 775-7. doi: 10.12968/denu.2013.40.9.770. PMID 24386769
- [Background] Burden DJ, Mullally BH, Robinson SN. Palatally ectopic canines: closed eruption versus open eruption. Am J Orthod Dentofacial Orthop. 1999 Jun;115(6):640-4. doi: 10.1016/s0889-5406(99)70289-1. PMID 10358246
- [Background] Parkin N, Benson PE, Thind B, Shah A. Open versus closed surgical exposure of canine teeth that are displaced in the roof of the mouth. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006966. doi: 10.1002/14651858.CD006966.pub2. PMID 18843740
- [Background] Wisth PJ, Norderval K, Booe OE. Comparison of two surgical methods in combined surgical-orthodontic correction of impacted maxillary canines. Acta Odontol Scand. 1976;34(1):53-7. doi: 10.3109/00016357609026558. PMID 1066949
- [Background] Gharaibeh TM, Al-Nimri KS. Postoperative pain after surgical exposure of palatally impacted canines: closed-eruption versus open-eruption, a prospective randomized study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Sep;106(3):339-42. doi: 10.1016/j.tripleo.2007.12.025. Epub 2008 Jun 11. PMID 18547839
- [Background] Parkin NA, Deery C, Smith AM, Tinsley D, Sandler J, Benson PE. No difference in surgical outcomes between open and closed exposure of palatally displaced maxillary canines. J Oral Maxillofac Surg. 2012 Sep;70(9):2026-34. doi: 10.1016/j.joms.2012.02.028. Epub 2012 Jun 6. PMID 22677328
- [Background] Chaushu S, Becker A, Zeltser R, Branski S, Vasker N, Chaushu G. Patients perception of recovery after exposure of impacted teeth: a comparison of closed- versus open-eruption techniques. J Oral Maxillofac Surg. 2005 Mar;63(3):323-9. doi: 10.1016/j.joms.2004.11.007. PMID 15742281
- [Background] Caminiti MF, Sandor GK, Giambattistini C, Tompson B. Outcomes of the surgical exposure, bonding and eruption of 82 impacted maxillary canines. J Can Dent Assoc. 1998 Sep;64(8):572-4, 576-9. PMID 9785687
- [Background] Wisth PJ, Norderval K, Boe OE. Periodontal status of orthodontically treated impacted maxillary canines. Angle Orthod. 1976 Jan;46(1):69-76. doi: 10.1043/0003-3219(1976)0462.0.CO;2. PMID 1062179
- [Background] Becker A, Kohavi D, Zilberman Y. Periodontal status following the alignment of palatally impacted canine teeth. Am J Orthod. 1983 Oct;84(4):332-6. doi: 10.1016/s0002-9416(83)90349-4. PMID 6578683
- [Background] Kohavi D, Becker A, Zilberman Y. Surgical exposure, orthodontic movement, and final tooth position as factors in periodontal breakdown of treated palatally impacted canines. Am J Orthod. 1984 Jan;85(1):72-7. doi: 10.1016/0002-9416(84)90124-6. PMID 6581728
- [Background] Schmidt AD, Kokich VG. Periodontal response to early uncovering, autonomous eruption, and orthodontic alignment of palatally impacted maxillary canines. Am J Orthod Dentofacial Orthop. 2007 Apr;131(4):449-55. doi: 10.1016/j.ajodo.2006.04.028. PMID 17418710
- [Background] Parkin NA, Milner RS, Deery C, Tinsley D, Smith AM, Germain P, Freeman JV, Bell SJ, Benson PE. Periodontal health of palatally displaced canines treated with open or closed surgical technique: a multicenter, randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):176-84. doi: 10.1016/j.ajodo.2013.03.016. PMID 23910198
- [Background] Zasciurinskiene E, Bjerklin K, Smailiene D, Sidlauskas A, Puisys A. Initial vertical and horizontal position of palatally impacted maxillary canine and effect on periodontal status following surgical-orthodontic treatment. Angle Orthod. 2008 Mar;78(2):275-80. doi: 10.2319/010907-8.1. PMID 18251594
- [Background] Quirynen M, Op Heij DG, Adriansens A, Opdebeeck HM, van Steenberghe D. Periodontal health of orthodontically extruded impacted teeth. A split-mouth, long-term clinical evaluation. J Periodontol. 2000 Nov;71(11):1708-14. doi: 10.1902/jop.2000.71.11.1708. PMID 11128918
- [Background] Smailiene D, Kavaliauskiene A, Pacauskiene I, Zasciurinskiene E, Bjerklin K. Palatally impacted maxillary canines: choice of surgical-orthodontic treatment method does not influence post-treatment periodontal status. A controlled prospective study. Eur J Orthod. 2013 Dec;35(6):803-10. doi: 10.1093/ejo/cjs102. Epub 2013 Jan 24. PMID 23349422
- [Background] Crescini A, Nieri M, Buti J, Baccetti T, Mauro S, Prato GP. Short- and long-term periodontal evaluation of impacted canines treated with a closed surgical-orthodontic approach. J Clin Periodontol. 2007 Mar;34(3):232-42. doi: 10.1111/j.1600-051X.2006.01042.x. Epub 2007 Jan 25. PMID 17257160
- [Background] Caprioglio A, Vanni A, Bolamperti L. Long-term periodontal response to orthodontic treatment of palatally impacted maxillary canines. Eur J Orthod. 2013 Jun;35(3):323-8. doi: 10.1093/ejo/cjs020. Epub 2012 Apr 24. PMID 22531665
- [Background] Powell CV, Kelly AM, Williams A. Determining the minimum clinically significant difference in visual analog pain score for children. Ann Emerg Med. 2001 Jan;37(1):28-31. doi: 10.1067/mem.2001.111517. PMID 11145767
- [Background] Bird SB, Dickson EW. Clinically significant changes in pain along the visual analog scale. Ann Emerg Med. 2001 Dec;38(6):639-43. doi: 10.1067/mem.2001.118012. PMID 11719742
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Parkin NA, Freeman JV, Deery C, Benson PE. Esthetic judgments of palatally displaced canines 3 months postdebond after surgical exposure with either a closed or an open technique. Am J Orthod Dentofacial Orthop. 2015 Feb;147(2):173-81. doi: 10.1016/j.ajodo.2014.10.026. PMID 25636550
- [Background] Ericson S, Kurol J. Early treatment of palatally erupting maxillary canines by extraction of the primary canines. Eur J Orthod. 1988 Nov;10(4):283-95. doi: 10.1093/ejo/10.4.283. No abstract available. PMID 3208843
- [Background] Fleming PS, Scott P, Heidari N, Dibiase AT. Influence of radiographic position of ectopic canines on the duration of orthodontic treatment. Angle Orthod. 2009 May;79(3):442-6. doi: 10.2319/042708-238.1. PMID 19413390
- [Background] Naoumova J, Kjellberg H. The use of panoramic radiographs to decide when interceptive extraction is beneficial in children with palatally displaced canines based on a randomized clinical trial. Eur J Orthod. 2018 Nov 30;40(6):565-574. doi: 10.1093/ejo/cjy002. PMID 29462471
- [Background] Bjorksved M, Arnrup K, Lindsten R, Magnusson A, Sundell AL, Gustafsson A, Bazargani F. Closed vs open surgical exposure of palatally displaced canines: surgery time, postoperative complications, and patients' perceptions: a multicentre, randomized, controlled trial. Eur J Orthod. 2018 Nov 30;40(6):626-635. doi: 10.1093/ejo/cjy070. PMID 30321323
- [Background] Ferguson DJ, Rossais DA, Wilcko MT, Makki L, Stapelberg R. Forced-eruption time for palatally impacted canines treated with and without ostectomy-decortication technique. Angle Orthod. 2019 Sep;89(5):697-704. doi: 10.2319/111418-809.1. Epub 2019 Mar 19. PMID 30888841
- [Background] Alqerban A, Jacobs R, Fieuws S, Willems G. Comparison of two cone beam computed tomographic systems versus panoramic imaging for localization of impacted maxillary canines and detection of root resorption. Eur J Orthod. 2011 Feb;33(1):93-102. doi: 10.1093/ejo/cjq034. PMID 21270321
- [Derived] Faerovig LF, Bjornland T, Magnusson A, Lindsten R, Pandis N, Bjerklin K, Vandevska-Radunovic V. Closed vs open surgical exposure of palatally displaced canines: Patients' perceptions of recovery, operating time, and complications-A 2-center randomized controlled trial. Am J Orthod Dentofacial Orthop. 2025 Apr;167(4):382-398. doi: 10.1016/j.ajodo.2024.11.014. PMID 40157786